CLINICAL TRIAL: NCT03678181
Title: Increasing Engagement and Improving HIV Care Outcomes Via Stigma Reduction in an Online Social Networking Intervention Among Racially Diverse Young Men Who Have Sex With Men and Transgender Women
Brief Title: Increasing Engagement and Improving HIV Outcomes Via HealthMPowerment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of North Carolina (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MD013623 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases; Stigma, Social
Keywords: Prevention; Internet; Adolescence; LGBT; Sexuality; Young Adulthood
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Social Stigma; Sexuality | interventions — HIV Testing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Information-Only Arm (Active Comparator): The HMP 2.0 Information-Only Control Arm will feature a streamlined version of the website that provides tailored information and content for YBLMT. This follows the design of HMP 1.0 where control arm participants had access to HIV-related Knowledge Center articles of the main intervention without access to the engagement features, interactive forums, or doctor Q&A. HIV-negative and sero-unknown participants also will be able to request HIV home test kits. The choice of control arm balances equipoise with research study design; in HMP 1.0, control arm participants also experienced a statistically significant intervention benefit.
  Interventions: Behavioral: Information Resources; Behavioral: HIV Testing
- HMP 2.0 Arm (Experimental): Participants in this experimental arm will receive access to HMP 2.0, an interactive site that includes a Knowledge Center focused on HIV prevention content, interactive forums, and a provider question & answer platform.
  Interventions: Behavioral: Information Resources; Behavioral: Social Support; Behavioral: HIV Testing
- Peer-referred HMP network arm (Experimental): Participants randomized to Intervention Arm 2 (peer-created network) will be enrolled into a parallel (but separate) version of HMP 2.0. The only difference between the two intervention arms is that the peer-referred HMP network arm will allow participants to refer and enroll 2 peers of their choosing into the study.
  Interventions: Behavioral: Information Resources; Behavioral: Social Support; Behavioral: HIV Testing

INTERVENTIONS:
Behavioral: Information Resources — The investigators will provide a HIV-related content as the attention-control condition.
Behavioral: Social Support — The investigators will provide evidence-based answers to users' health questions, including linkage to care.
  Arms: HMP 2.0 Arm; Peer-referred HMP network arm
Behavioral: HIV Testing — The investigators will provide opportunities for participants to get tested through HIV home test kits.

SUMMARY:
The overall goal of this 3-arm randomized trial is to test whether a network-driven online intervention tailored for intersectional stigma amelioration can elicit online social support, promote intervention engagement, and mitigate the impact of multiple stigmas on HIV-related outcomes among young Black and/or Latino men who have sex with men and transgender women.

DETAILED DESCRIPTION:
Multiple stigmas related to sexuality, race, and HIV infection negatively impact HIV testing, engagement in HIV care, and consistent viral suppression (VS) among young Black or Latino men who have sex with men and transgender women (YBLMT). At present, few interventions have addressed the effects of intersectional stigma among people living with HIV and HIV affected populations. This study tests whether an online intervention tailored for intersectional stigma amelioration can elicit online social support, promote intervention engagement, and mitigate the impact of multiple stigmas on HIV-related outcomes. This study will recruit and enroll 1,050 young (ages 15-29), racially and ethnically diverse men who have sex with men and transgender women affected by HIV across the United States. Using a HIV-status stratified randomized trial design, participants will be assigned into one of three conditions (information-only control, a researcher-driven social network intervention, or a peer-driven social network intervention). Behavioral assessments will occur at baseline, 3, 6, 9 and 12 months; biomarkers (viral load) are scheduled for baseline, 6 and 12 months. The primary outcome is stratified by HIV status and defined as successful engagement in care (consistent VS for HIV-positive participants and routine testing for HIV-negative participants). The specific aims are: 1) Test whether an online intervention that promotes user-generated content and engagement to address intersectional stigma is associated with improvements in the HIV prevention and care continuum (HIV testing, antiretroviral adherence, VS) as compared to an information-only control arm; 2) Explore whether user engagement, as measured by quantitative and qualitative paradata, mediates the intervention's stigma- and HIV care-related outcomes; and, 3) Examine how changes in intersectional stigma and improvements across the HIV care continuum vary between the researcher-driven vs. peer-driven social network intervention conditions. The research study is innovative given its focus on intersectional stigma as a key target of intervention, and its ability to assess how different kinds of online social network structures influence participants' engagement over time, reduce experiences of intersectional stigma, and improve successful engagement in care. This research addresses a critical need to reduce the effects of multiple stigmas in a priority population using an intervention delivered through a highly appealing, widely-utilized technology. If effective, this form of stigma amelioration via online support can be broadly disseminated to reduce HIV transmission and improve care among YBLMT.

ELIGIBILITY:
Inclusion Criteria:

* Ages 15-29 (inclusive);
* Identify as Black/African American and/or Latino/Hispanic;
* Be U.S. residents (verified by zip code);
* Report at least one episode of condomless anal sex act with a man in prior 6 months;
* Assigned male sex at birth;
* Currently identifies as male or as woman
* Have access to internet
* Reports owning or having regular access to a smartphone device or laptop/tablet through which to log onto the study site.

Exclusion Criteria:

* Assigned female sex at birth
* Aged 14 years or younger or 30 years or older at time of screening
* Does not speak or read English or Spanish
* Did not have consensual anal sex with a male partner in the prior 6 months
* Does not reside in the United States
* Currently incarcerated
* Planning to move out of the United States in next 12 months

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender men and transgender women are eligible.
Enrollment: 750 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Muessig, PhD, Principal Investigator — University of North Carolina; Jose A Bauermeister, PhD, Principal Investigator — University of Pennsylvania; Lisa Hightow-Weidman, MD, Study Director — University of North Carolina
Locations (3):
- United States (3):
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
The investigators will assure the timely release and sharing of data two years after the publication of the main trial findings from the final dataset. Study variables will be available; however, the investigators will protect the rights and privacy of human subjects by redacting all identifiers from the dataset. The de-identified data from this project will be available through individual requests directed to the Principal Investigators.

REFERENCES:
- [Derived] Muessig KE, Golinkoff JM, Hightow-Weidman LB, Rochelle AE, Mulawa MI, Hirshfield S, Rosengren AL, Aryal S, Buckner N, Wilson MS, Watson DL, Houang S, Bauermeister JA. Increasing HIV Testing and Viral Suppression via Stigma Reduction in a Social Networking Mobile Health Intervention Among Black and Latinx Young Men and Transgender Women Who Have Sex With Men (HealthMpowerment): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Dec 16;9(12):e24043. doi: 10.2196/24043. PMID 33325838

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Information-Only Arm | HMP 2.0 Arm | Peer-referred HMP Network Arm
Started | 332 | 333 | 85
Completed | 332 | 333 | 85
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Information-Only Arm | HMP 2.0 Arm | Peer-referred HMP Network Arm | Total
Number analyzed (Participants) | 332 | 333 | 85 | 750
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.72 (3.20) | 24.62 (3.52) | 26.18 (2.77) | 24.84 (3.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 332 | 333 | 85 | 750
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 140 | 152 | 26 | 318
  Not Hispanic or Latino | 192 | 181 | 59 | 432
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 5 | 0 | 12
  Asian | 2 | 3 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 208 | 181 | 64 | 453
  White | 20 | 40 | 5 | 65
  More than one race | 32 | 29 | 7 | 68
  Unknown or Not Reported | 63 | 74 | 8 | 145
HIV Status [Count of Participants; unit: Participants] — Participant self-reported HIV status
  Participants
    HIV negative | 258 | 258 | 4 | 520
    HIV positive | 74 | 75 | 81 | 230

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Reporting Changes in Their HIV Testing Behavior Using Self-report Questionnaires
Description: The investigators will estimate the proportion of participants who test at least twice for HIV over a 12-month period by intervention group.
Time Frame: 12 month
Population: HIV Testing outcome focuses on HIV-negative participants in the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Information-Only Arm | HMP 2.0 Arm | Peer-referred HMP Network Arm
Number analyzed (Participants) | 258 | 258 | 4
Participants | 185 | 171 | 2

2. Primary Outcome: Percent of Participants Reporting Viral Suppression Using Self-Report Questionnaires
Description: The investigators will estimate the proportion of participants living with HIV who achieve viral suppression over a 12-month period by intervention group.
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Information-Only Arm | HMP 2.0 Arm | Peer-referred HMP Network Arm
Number analyzed (Participants) | 74 | 75 | 81
Participants
  Virally Suppressed | 45 | 60 | 60
  Not Virally Suppressed | 29 | 15 | 21

3. Secondary Outcome: Number of Days in the Prior Week That Participants Self-report Missing at Least One Dose of Their Adherence to Antiretroviral Therapy (ART) Using a Self-Reported Questionnaire
Description: The investigators will test the proportion of the HIV-positive sample that adheres to their HIV care regimen during the 12-month follow-up.
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Information-Only Arm | HMP 2.0 Arm | Peer-referred HMP Network Arm
Number analyzed (Participants) | 40 | 53 | 51
days | 0.92 (1.65) | 0.96 (1.75) | 1.21 (2.06)

4. Secondary Outcome: Percent of Participants Reporting PrEP Uptake Using Self-Report Questionnaires
Description: The investigators will test the proportion of the HIV-negative sample that reports using PrEP by the 12-month follow-up.
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Information-Only Arm | HMP 2.0 Arm | Peer-referred HMP Network Arm
Number analyzed (Participants) | 205 | 189 | 2
Participants
  Yes, I am on PrEP right now | 77 | 74 | 0
  Yes, I was in the past, but I'm not on PrEP anymore | 50 | 42 | 1
  No, I've never taken PrEP | 78 | 73 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the year of study participation.
Arm/Group | Information-Only Arm | HMP 2.0 Arm | Peer-referred HMP Network Arm
All-Cause Mortality (participants affected / at risk) | 0/332 | 0/333 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/332 | 0/333 | 0/85
Other Adverse Events (participants affected / at risk) | 0/332 | 0/333 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03678181/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03678181/ICF_001.pdf